CLINICAL TRIAL: NCT02769429
Title: Is There a Difference Between Posterior Approach Ultrasound-guided Continuous Interscalene Block (Upper Trunk Block) and Stimulator Guided Continuous Cervical Paravertebral Block (C6 Root Block)?
Brief Title: Continuous Blockade of the Brachial Plexus
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: I. Heermann Anesthesia Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB201600012
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Arthroses; Degenerative Disorder; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ultrasound-guided CISB: Group 1 will receive ultrasound-guided CISB with the catheter placed on the upper trunk of the brachial plexus
  Interventions: Device: Ultrasound-guided CISB
- nerve stimulator-guided CCPVB: Group 2 will receive landmark with nerve stimulator based needle placement and then nerve stimulator-guided CCPVB with the catheter placed on the 6th cervical spinal root
  Interventions: Device: nerve stimulator-guided CCPVB

INTERVENTIONS:
Device: Ultrasound-guided CISB — This group will receive ultrasound-guided CISB with the catheter placed on the upper trunk of the brachial plexus
  Groups: ultrasound-guided CISB
Device: nerve stimulator-guided CCPVB — This group will receive landmark with nerve stimulator based needle placement and then nerve stimulator-guided CCPVB with the catheter placed on the 6th cervical spinal root
  Groups: nerve stimulator-guided CCPVB

SUMMARY:
This study will answer the question whether there is a difference in the effects and complication rates of ultrasound guided continuous interscalene block (CISB) and nerve stimulation-guided continuous cervical paravertebral block (CCPVB). The aim of this study is to evaluate the differences in efficacy and side effects - if any.

DETAILED DESCRIPTION:
This is a prospective randomized double-blinded study that will compare two commonly used approaches for the continuous blockade of the brachial plexus: the CCPVB, which focusses on the six cervical nerve root (C6 root), and CISB, which focuses on the upper trunk of the brachial plexus. Data of sensory testing, motor strength, shoulder pain, phrenic nerve function, recurrent laryngeal nerve (RNL) function, ipsilateral Horner's syndrome, block time and medication doses used for block placement, will be collected. All observations and measurements will be made by a member of the research team who is unaware of patient allocation to any particular group.

ELIGIBILITY:
Inclusion Criteria:

* The general inclusion will be those adult patients who:

  * are between the ages of 18 and 80 years
  * have an ASA Health Classification of I, II, or III
  * are scheduled for shoulder arthroplasty or rotator cuff repair surgery
  * Patients with a BMI of =to/< 40 Exclusion

The Exclusion criteria will include:

* Patient refusal to participate in the study or sign informed consent
* Patients with contraindications to any of the two blocks or allergy to any of the drugs used
* Patients with shoulder surgery that developed into any other surgery other than total shoulder arthroplasty or rotator cuff repair
* Patients with a BMI >40

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are are scheduled for shoulder arthroplasty or rotator cuff repair surgery at an area hospital
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Changes between the two groups assessed by sensory testing | Change from baseline up to 7 days (end of catheter placement)
  Sensory abnormalities will be assessed by sensation of cold and dermatomes sensation.

SECONDARY OUTCOMES:
Changes between the two groups assessed by motor strength | Change from baseline up to 7 days (end of catheter placement)
  Motor strength will be assessed on a scale of 0 to 5 Medical Research Council (MRC) scale
Changes between the two groups assessed by shoulder pain | Change from baseline up to 7 days (end of catheter placement)
  Shoulder pain will be assessed by the Defense and Veterans Pain Rating Scale (DVPRS) where pain will be rated as no pain, mild, moderate, or severe pain, and on a scale of 0 to 10 where 0 represents no pain, 1 to 3 represents mild pain, 4 to 6 represents moderate pain, 7 to 9 represents severe pain, and 10 represents the worst pain imaginable where nothing else but the pain matters
Changes between the two groups assessed by Phrenic nerve function | Change from baseline up to 7 days (end of catheter placement)
  Phrenic nerve function will be evaluated by measuring the movements of the diaphragm by ultrasonography or the inability to visualize using ultrasound (US)
Changes between the two groups assessed by recurrent laryngeal nerve (RLN) function | Change from baseline up to 7 days (end of catheter placement)
  RLN function will be assessed by hoarseness or swallowing difficulty
Changes between the two groups assessed by development of ipsilateral Horner's syndrome | Change from baseline up to 7 days (end of catheter placement)
  Development of ipsilateral Horner's syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Yury Zasimovich, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Florida Surgical Center, Gainesville, Florida
  - UF Health, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No